# STATISTICAL ANALYSIS PLAN (SAP)

**Study:** Levetiracetam Versus Phenobarbitone for the Treatment of Neonatal Seizures in a

Tertiary Care Hospital

Principal Investigator: Dr. Gohar Ali

| Official Study Title: |
|---|
| Levetiracetam Versus Phenobarbitone for the Treatment of Neonatal Seizures in a |
| Tertiary Care Hospital |
| Short title/acronyms: Levetiracetam Versus Phenobarbitone for the Treatment of Neonatal |
| Seizures |
| ClinicalTrials.gov Identifier: |
| NCT Not Yet Assigned |
| Organization's Unique Protocol ID: |
| DHQ-DIK-IREB NO. 4806 |
| Document Type: |
| Statistical Analysis Plan (SAP) |
| Date: |
| Study Start Date |
| April 08 2024 |
| Primary Completion Date |
| March 31 2025 |
| Study Completion Date |
| April 10 2025 |
| Prepared By: |
| Dr. Gohar Ali |

#### **Analysis Population**

- All randomized neonates (Intention-to-Treat, ITT)
- **Per-protocol population** for sensitivity analysis (neonates who completed treatment as per protocol)

### **Descriptive Statistics**

- Continuous variables: mean  $\pm$  SD or median (IQR)
- Categorical variables: frequency (%)

#### **Outcome Analysis**

### **Primary Outcome:**

- •Seizure control rate within 24 hours
- Compare seizure control between levetiracetam and phenobarbitone groups
- Statistical Test: Chi-square or Fisher's exact test
- Significance level:  $\alpha = 0.05$

#### **Secondary Outcome Analysis**

- Time to seizure cessation
  - Independent t-test or Mann–Whitney U test
- Need for second-line anticonvulsant
  - Chi-square test
- Seizure recurrence during hospital stay
  - Chi-square test
- Adverse drug reactions
  - Chi-square test
- Mortality during hospital stay
  - Chi-square test

## **Subgroup Analysis (optional)**

- Preterm vs Term neonates
- Birth weight  $<2500 \text{ g vs} \ge 2500 \text{ g}$
- Etiology of seizures (HIE vs metabolic vs infection vs others)

## **Handling Missing Data**

- Multiple imputation if missing data > 5%
- Sensitivity analysis comparing complete case vs imputed dataset

#### **Software**

• Analysis performed using SPSS version 23,

## Reporting

- Two-sided p-values
- 95% confidence intervals for effect estimates
- Tables and figures for primary and secondary outcomes